CLINICAL TRIAL: NCT05692089
Title: Incidence of Infective Endocarditis in End Stage Renal Disease Patients on Hemodialysis by Transesophageal Echocardiography in Assuit University Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christin Nashaat Sedeek Aziz, Resident Doctor, Assiut University
Other Study IDs: Infective endocarditis in ESRD
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Infective Endocarditis; End Stage Renal Disease
MeSH Terms: conditions — Endocarditis; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
1. To detect in more detail the incidence of infective endocarditis in patients with end stage renal disease (ESRD) on hemodialysis.
2. To compare the relationship between different forms of haemodialysis access type and the related incidence of infective endocarditis.
3. To determine individual risk factors, including type of vascular haemodialysis access, previous valve lesion and immunocompromised patients.

DETAILED DESCRIPTION:
All patients will undergo TTE and TEE within 36 hours of symptoms. TTE will be performed with a 2.5- or 3.5-MHz phased-array transducer. Patients will fast for more than 4 hours before TEE, which will be performed under local pharyngeal anesthesia; the majority of patients will also receive intravenous midazolam (0.5 to 2.0 mg). A 5-MHz phased-array transducer (either biplane or multiplane) will be used for the transesophageal examination, which consisted principally of two-dimensional imaging and color flow mapping and will be performed without any complications in all patients.

All echocardiograms will be evaluated later during reading sessions by two observers. TTE studies will be defined as technically inadequate if both observers deemed the quality of the images to be insufficient to gain diagnostic information regarding the presence or absence of vegetations or their complications. Findings on TTE and TEE will be separately categorized as indicating high, intermediate, or low probability for endocarditis as follows: high, any definite vegetation and/or abscess or probable vegetation with evidence of otherwise unexplained valvular dysfunction (greater than mild regurgitation or a paravalvular prosthetic leak); intermediate, a probable vegetation without evidence of unexplained valvular dysfunction; and low, no evidence of vegetation or abscess or a possible vegetation without any evidence of regurgitation. 3 sets of blood culture with one hour interval will be withdrawn from the central line from all patients, before stating antibiotics within 24 hours from the onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Incidence of infective endocarditis in ESRD that on hemodialysis.
* Must be fit for Transoesophageal ECHO.

Exclusion Criteria:

* Any patient with sepsis due to causes other than infected vascular access.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Statistical tests: Categorical variables will be expressed as a frequency and a percentage and compared with the chi-square test and the Fisher exact test when necessary. Quantitative variables will be expressed as median and interquartile range or mean and standard deviation. Assessment of normality and equality of variances for continuous data will be performed using the Shapiro-Wilk test and the Levene test, respectively. Thereafter, continuous variables will be compared by a Student t-test, Mann-Whitney U test or Fisher-Pitman permutation test as necessary. Multivariable Cox regression was fitted to examine the dependence of infective endocarditis on RRTs (haemodialysis, CVC [external or tunnelled], arteriovenous fistula, arteriovenous graft, and kidney transplantation).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of infective endocarditis in end stage renal disease patients on hemodialysis | Baseline
  by transesophageal echocardiography in Assiut university hospital. The endpoint was infective endocarditis diagnosed according to Dukes criteria for diagnosis of infective endocarditis (Roidad et al.,2010) by transthoracic or transesophageal echocardiography and positive repeated blood cultures.

SECONDARY OUTCOMES:
Infective endocarditis complications | Baseline
  Secondary (subsidiary): Patients presented by infective endocarditis complications such as refractory heart failure, distal embolization, cerebral haemorrhage, pyrexia of unknown origin.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mohammed Ali, PhD, Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine-Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudry MS, Carlson N, Gislason GH, Kamper AL, Rix M, Fowler VG Jr, Torp-Pedersen C, Bruun NE. Risk of Infective Endocarditis in Patients with End Stage Renal Disease. Clin J Am Soc Nephrol. 2017 Nov 7;12(11):1814-1822. doi: 10.2215/CJN.02320317. Epub 2017 Oct 3. PMID 28974524
- [Background] Iung B, Rouzet F, Brochet E, Duval X. Cardiac Imaging of Infective Endocarditis, Echo and Beyond. Curr Infect Dis Rep. 2017 Feb;19(2):8. doi: 10.1007/s11908-017-0560-2. PMID 28233189
- [Background] Bruun NE, Habib G, Thuny F, Sogaard P. Cardiac imaging in infectious endocarditis. Eur Heart J. 2014 Mar;35(10):624-32. doi: 10.1093/eurheartj/eht274. Epub 2013 Jul 30. PMID 23900698
- [Background] McCarthy JT, Steckelberg JM. Infective endocarditis in patients receiving long-term hemodialysis. Mayo Clin Proc. 2000 Oct;75(10):1008-14. doi: 10.4065/75.10.1008. PMID 11040848
- [Background] Stevenson KB, Adcox MJ, Mallea MC, Narasimhan N, Wagnild JP. Standardized surveillance of hemodialysis vascular access infections: 18-month experience at an outpatient, multifacility hemodialysis center. Infect Control Hosp Epidemiol. 2000 Mar;21(3):200-3. doi: 10.1086/501744. PMID 10738990
- [Background] Roidad N, Rhodes L, Warden B. A review of the American Heart Association revised guidelines for the prevention of infective endocarditis. W V Med J. 2010 May-Jun;106(3):12-5. No abstract available. PMID 21736149